CLINICAL TRIAL: NCT06520540
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Multiple Oral Administration of HDM1002 Tablets in Chinese Overweight and Obese Adult Subjects
Brief Title: HDM1002 Tablets in Chinese Overweight and Obese Adult Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDM1002-103
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Glucagon-Like Peptide-1 Receptor Agonists
Keywords: Glucagon-Like Peptide-1 Receptor Agonists; HDM1002 tablet; Chinese overweight and obese adult

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HDM1002 100 mg (Active Comparator)
  Interventions: Drug: HDM1002 100 mg QD 12weeks; Drug: HDM1002 200 mg QD 12weeks; Drug: HDM1002 400 mg QD 12weeks，Q 2W for titration; Drug: HDM1002 400 mg QD 12weeks，Q 3W for titration
- HDM1002 200 mg (Active Comparator)
  Interventions: Drug: HDM1002 200 mg QD 12weeks; Drug: HDM1002 400 mg QD 12weeks，Q 2W for titration; Drug: HDM1002 400 mg QD 12weeks，Q 3W for titration
- HDM1002 400 mg (Active Comparator)
  Interventions: Drug: HDM1002 400 mg QD 12weeks，Q 2W for titration; Drug: HDM1002 400 mg QD 12weeks，Q 3W for titration
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Drug: HDM1002 100 mg QD 12weeks — Participants received maintenance dose of 100 mg HDM1002 administered orally once daily (QD)
  Arms: HDM1002 100 mg
Drug: HDM1002 200 mg QD 12weeks — Participants received maintenance dose of 200 mg HDM1002 administered orally once daily (QD)
  Arms: HDM1002 100 mg; HDM1002 200 mg
Drug: HDM1002 400 mg QD 12weeks，Q 2W for titration — Participants received maintenance dose of 400 mg HDM1002 administered orally once daily (QD) Q 2W for titration
  Arms: HDM1002 100 mg; HDM1002 200 mg; HDM1002 400 mg
Drug: HDM1002 400 mg QD 12weeks，Q 3W for titration — Participants received maintenance dose of 400 mg HDM1002 administered orally once daily (QD) Q 3W for titration
  Arms: HDM1002 100 mg; HDM1002 200 mg; HDM1002 400 mg
Device: Placebo — Placebo
  Arms: Placebo

SUMMARY:
• To assess the safety of multiple oral doses of HDM1002 tablets under different titrations in Chinese overweight and obese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese subjects aged 18 to 60 years (including 18 years and 60 years old), either male or female subjects;
2. BMI at 24.0 to 36.0 kg at screening and at random / m2Between (including 24.0 and 36.0 kg / m2）；
3. For fertile subjects, female subjects from 14 days before the informed consent form (ICF) to 30 days after the last administration, male subjects within 90 days after the ICF to the last administration, without birth planning and agreed to highly effective contraception (see Section 5.2.3 for details);
4. Ability to understand the procedures and methods of this study, voluntarily sign the ICF, and be willing to strictly comply with the clinical trial protocol requirements to complete the relevant process.

Exclusion Criteria:

Selection criteria:

Subjects must meet all of the following inclusion criteria to be enrolled in this study:

1. Chinese subjects aged 18 to 60 years (including 18 years and 60 years old), either male or female subjects;
2. BMI at 24.0 to 36.0 kg at screening and at random / m2Between (including 24.0 and 36.0 kg / m2）；
3. For fertile subjects, female subjects from 14 days before the informed consent form (ICF) to 30 days after the last administration, male subjects within 90 days after the ICF to the last administration, without birth planning and agreed to highly effective contraception (see Section 5.2.3 for details);
4. Ability to understand the procedures and methods of this study, voluntarily sign the ICF, and be willing to strictly comply with the clinical trial protocol requirements to complete the relevant process.

Exclusion criteria:

Subjects meeting either of the following criteria will be excluded:

1. 5% self-reported or documented body weight change within 3 months prior to randomization;
2. Previous diagnosis of type 1, type 2 or any other type of diabetes; or using hypoglycemic drugs; or HbA1c 6.5% at screening or fasting glucose 7.0 mmol/L; or fasting glucose <3.9 mmol / L;
3. Diagnosis of overweight or obesity caused by other diseases or drugs;
4. History or family history of medullary thyroid carcinoma, thyroid C cell hyperplasia, or multiple endocrine adenomatosis type 2;
5. History of chronic pancreatitis or onset of acute pancreatitis within 3 months before signing an ICF;
6. History of acute gallbladder disease within 3 months before signing the ICF;
7. Any malignant tumor within 5 years before signing the ICF (except for basal cell carcinoma that has received curative treatment and is considered cured);
8. Combination of cardiovascular and cerebrovascular diseases with obvious clinical significance, including but not limited to angina pectoris, MI, stroke or severe peripheral artery circulation disorder within 1 year before signing ICF; presence of risk factors of torsade ventricular tachycardia; presence of untreated serious arrhythmia, such as sick sinus syndrome, second or third degree atrioventricular block; or screening systolic blood pressure 160 mmHg, or diastolic blood pressure 100 mmHg;
9. In the judgment of the investigator, the subjects had some diseases or conditions that may affect drug absorption, such as active inflammatory bowel disease, gastrectomy resection, any intestinal area resection, etc.;
10. Those who had major surgery within 3 months prior to signing the ICF or who performed surgery during the planned study;
11. According to the investigator, the presence of concomitant diseases, including but not limited to the respiratory system, digestive system, nervous system, urogenital system, blood system, endocrine system and other diseases;
12. Known intolerance or hypersensitivity to a GLP-1 receptor (GLP-1R) agonist;
13. Within 3 months prior to ICF signing, the following drugs were used and significantly weight, including but not limited to: a. Drugs or products with weight loss effects, such as GLP-1R agonists (liraglutide, selmeaglutide, benallutide, etc.), orlistat, naltrexone / bupropion, etc.; b. Drugs or products that increase body weight, such as systemic corticosteroids, psychiatric medication (e. g., tricyclic antidepressants, paroxetine, olanzapine, clozapine, mirtazapine, valproic acid and its derivatives, etc.); c. Any Chinese patent medicine or Chinese herbal medicine that may affect the body weight;
14. Any drug used within 14 days or may affect the pharmacokinetics of HDM1002 tablets (whichever is older) (see Section 6.4.2 and Section 6.4.3), including prescription drugs, over-the-counter drugs, Chinese herbal medicines, proprietary Chinese medicines, or nutritional supplements;
15. Subjects taking lipid-lowering drugs within 30 days before signing ICF;
16. Have participated in any clinical trial within 30 days before randomization or within 5 half-lives after the last dose (whichever is older) (except for signed ICF with no drug or device intervention);
17. Any of the laboratory indicators during the screening period met the following criteria:

    1. <110 g / L for women and <120 g / L for men;
    2. glutamate aminotransferase> 2.0 upper limit of normal (ULN), or aminotransferase> 2.0 ULN, or alkaline phosphatase> 1.5 x ULN, or total bilirubin> 1.5 ULN (subjects with Gil bert's syndrome can participate in this study with direct bilirubin ULN);
    3. Triglycerides> 5.6 mmol / L;
    4. Calcitonin: 35 ng/L;
    5. Thyroid-stimulating hormone> 6.0 mIU / L or <0.4 mIU / L;
    6. Blood amylase or lipase> ULN;
    7. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m, calculated from the Cooperative Epidemiological Study of Chronic Kidney Disease (CKD-EPI) formula2；
18. The following ECG abnormalities were present during the screening period: QTcF> 450 ms, or heart rate <50 beats / min or> 100 beats / min;
19. Positive test results for hepatitis B virus surface antigen, hepatitis C virus antibody or treponema pallidum antibody, or non-negative for human immunodeficiency virus;
20. More than 5 cigarettes per day in the 3 months before signing the ICF;
21. Those who had drunk alcohol abuse within 1 year before signing the ICF (i. e., drinking more than 14 standard units per week for men, women drinking more than 7 standard units per week, 1 standard unit containing 14 g alcohol, such as 360 ml beer or 150 ml alcohol of 40 ml), or prerandomized alcohol breath test or blood alcohol test positive;
22. History of addictive drug abuse within 1 year before signing the ICF, or positive urine drug test before randomization;
23. Within 7 days prior to randomization, subjects reported having consumed grapefruit or products containing grapefruit;
24. Pregnancy (blood human chorionic gonadotropin 5 mIU / ml or positive urine pregnancy test) or lactating women;
25. The subject is the investigator or other relevant investigator of the project;
26. In the opinion of the investigator, the subject was not fit to participate in any other condition of the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-28 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
TEAEs, SAEs, AEs leading to withdrawal, and AEs leading to death, AEs of special interest | Baseline, Week 12
  TEAEs and SAEs (incidence, severity and causal relationship), AEs leading to withdrawal, and AEs leading to death, AEs of special interest

SECONDARY OUTCOMES:
change in body weight from baseline at Day 85 | Baseline, Week 12
  Weight during treatment from baseline
change in BMI from baseline at Day 85 | Baseline, Week 12
  change in body mass index (BMI) from baseline
change in waist circumference from baseline at Day 85 | Baseline, Week 12
  Change in waist circumference from baseline
Plasma PK parameters | Baseline, Week 12
  Cmax
Plasma PK parameters | Baseline, Week 12
  Tmax
Plasma PK parameters | Baseline, Week 12
  AUC0-last
Plasma PK parameters | Baseline, Week 12
  AUCtau
Plasma PK parameters | Baseline, Week 12
  AUC0-24h
Plasma PK parameters | Baseline, Week 12
  AUC0-∞
Plasma PK parameters | Baseline, Week 12
  t1/2z
Plasma PK parameters | Baseline, Week 12
  CL/F
Plasma PK parameters | Baseline, Week 12
  Vz/F

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, Principal Investigator — Zhongshan Hospital, Shanghai, China
Locations (1):
- HDM1002, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No